CLINICAL TRIAL: NCT00041964
Title: A Prospective Observational Study of Virologic and Immunologic Changes in HIV-Infected Women During the Postpartum Period
Brief Title: A Study of HIV Levels During Pregnancy and After Childbirth
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5150; ACTG A5153s; AACTG A5150; AACTG A5153s
Record Dates: First submitted 2002-07-19; First posted 2002-07-22 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections; Pregnancy
Keywords: Lopinavir; Pregnancy Trimester, Third; Pregnancy Complications, Infectious; HIV Protease Inhibitors; Ritonavir; Nelfinavir; Viral Load; puerperium
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious

SUMMARY:
The purpose of this study is to find out if HIV-infected pregnant women taking anti-HIV drugs have an increased amount of HIV in their blood (viral load) after having the baby.

The purpose of A5153s, a substudy of A5150, is to characterize two anti-HIV drugs (nelfinavir [NFV] and lopinavir/ritonavir [LPV/r]) in HIV-infected women during pregnancy and after childbirth.

Sometimes pregnant women have an increase in their HIV viral load after their baby is born. This study will try to find out how often this happens. It will also examine possible reasons why the increase in viral load occurs.

DETAILED DESCRIPTION:
Limited data suggest that HIV-infected pregnant women develop postpartum viral rebound. However, viral load changes in the postpartum period have not been adequately characterized. Changes in adherence to antiretroviral therapy, pregnancy-related changes in pharmacokinetics of antiretroviral medications, and decline in immune competence are mechanisms by which postpartum viral load rebound may occur. This study is designed to characterize the incidence and magnitude of postpartum viral rebound during the initial 24 weeks postpartum and to explore the mechanisms and consequences of viral rebound.

Eligible patients are evaluated at gestational weeks 34 and 36, at delivery, and at regular visits for 96 weeks postpartum. Most evaluations include a medical history, physical exam, laboratory tests, and adherence and quality-of-life questionnaires. Viral load and CD4/CD8 cell counts are measured frequently.

Patients are expected to receive at least 8 weeks of stable HAART before delivery, and to continue HAART throughout the remainder of the study. The choice of HAART is left to the primary provider. No antiretroviral drugs are provided by this study.

Patients participating in the A5153s substudy receive either NFV or LPV/r as part of their HAART. Pharmacokinetic blood sampling takes place at 36 weeks gestation, 6 weeks postpartum, and 24 weeks postpartum. Patients record the administration times and doses of their NFV or LPV/r for 48 hours prior to each substudy visit, and hold their regularly scheduled doses of antiretroviral medications on substudy days. Patients arrive at the clinic fasting (no food or drink for the previous 8 hours) and are given a standardized breakfast prior to supervised administration of their NFV or LPV/r dose. An intravenous catheter is placed in an arm vein for blood collection at pre-dose and 1, 2, 4, and 6 hours post-dose.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are age 13 or older.
* Are between 22 and 30 weeks pregnant.
* Have had their pregnancy confirmed by ultrasound at 14 weeks gestation or later.
* Are infected with HIV.
* Are planning to receive at least 8 weeks of highly active antiretroviral therapy (HAART) by the time they have their baby.
* Are available for follow-up for the duration of the study.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Intend to terminate their pregnancy.
* Intend to breast-feed their baby.
* Are carrying a baby with major abnormalities, including spina bifida, anencephaly, hydrops, or ascites.
* Have taken certain medications.
* Are enrolled in other studies that require large blood draws.
* Will be taking anti-HIV drugs only to prevent mother-to-child transmission of HIV, and not to treat the maternal infection itself.
* Actively abuse drugs or alcohol in a way that would interfere with participation in the study.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Sha, Study Chair; Alice Stek, Study Chair
Locations (32):
- United States (31):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Los Angeles County Medical Center/USC, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - UCSD Mother, Child & Adolescent HIV Program, San Diego, California
  - San Francisco General Hosp, San Francisco, California
  - Univ of Florida- Health Science Ctr, Jacksonville, Florida
  - Emory Univ, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Cook County Hosp Core Ctr, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Chicago Childrens Memorial Hospital (Pediatric), Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Hutzel Hospital, Detroit, Michigan
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Hennepin County Med Clinic, Minneapolis, Minnesota
  - Univ of Med & Dentistry of NJ/Univ Hosp, Newark, New Jersey
  - NYU/Bellevue, New York, New York
  - Columbia University, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Jacobi Med Ctr, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Miriam Hosp / Brown Univ, Providence, Rhode Island
  - The Regional Med Ctr, Memphis, Memphis, Tennessee
  - Comprehensive Care Clinic, Nashville, Tennessee
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Univ of Washington (Seattle), Seattle, Washington
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Background] Melvin AJ, Burchett SK, Watts DH, Hitti J, Hughes JP, McLellan CL, King PD, Johnson EJ, Williams BL, Frenkel LM, Coombs RW. Effect of pregnancy and zidovudine therapy on viral load in HIV-1-infected women. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Mar 1;14(3):232-6. doi: 10.1097/00042560-199703010-00006. PMID 9117455
- [Background] Rich KC, Siegel JN, Jennings C, Rydman RJ, Landay AL. CD4+ lymphocytes in perinatal human immunodeficiency virus (HIV) infection: evidence for pregnancy-induced immune depression in uninfected and HIV-infected women. J Infect Dis. 1995 Nov;172(5):1221-7. doi: 10.1093/infdis/172.5.1221. PMID 7594657
- [Background] Cao Y, Krogstad P, Korber BT, Koup RA, Muldoon M, Macken C, Song JL, Jin Z, Zhao JQ, Clapp S, Chen IS, Ho DD, Ammann AJ. Maternal HIV-1 viral load and vertical transmission of infection: the Ariel Project for the prevention of HIV transmission from mother to infant. Nat Med. 1997 May;3(5):549-52. doi: 10.1038/nm0597-549. PMID 9142125
- [Background] Burns DN, Landesman S, Minkoff H, Wright DJ, Waters D, Mitchell RM, Rubinstein A, Willoughby A, Goedert JJ. The influence of pregnancy on human immunodeficiency virus type 1 infection: antepartum and postpartum changes in human immunodeficiency virus type 1 viral load. Am J Obstet Gynecol. 1998 Feb;178(2):355-9. doi: 10.1016/s0002-9378(98)80025-2. PMID 9500499
- [Result] Sha BE, Tierney C, Cohn SE, Sun X, Coombs RW, Frenkel LM, Kalams SA, Aweeka FT, Bastow B, Bardeguez A, Kmack A, Stek A; Aids Clinical Trials Group ACTG A5150 Team. Postpartum viral load rebound in HIV-1-infected women treated with highly active antiretroviral therapy: AIDS Clinical Trials Group Protocol A5150. HIV Clin Trials. 2011 Jan-Feb;12(1):9-23. doi: 10.1310/hct1201-9. PMID 21388937